CLINICAL TRIAL: NCT03111303
Title: Nosocomial Pneumonia as a Factor Influencing Parameters of Mechanical Ventilation: Results of a Retrospective, Observational Study
Brief Title: Mechanical Ventilation Parameters in HAP Patients
Status: Completed | Type: Observational
Sponsor: University Hospital Olomouc (Other)
Responsible Party: Principal Investigator, Radovan Uvizl, MD, Ph.D., University Hospital Olomouc
Other Study IDs: 65/16
Record Dates: First submitted 2017-04-07; First posted 2017-04-12 (Actual); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Mechanical Ventilation Pressure High
MeSH Terms: interventions — Respiration, Artificial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HAP patients: Mechanical ventilation, patients fulfilled HAP criteria
  Interventions: Device: mechanical ventilation
- non HAP patients: Mechanical ventilation, patients without HAP
  Interventions: Device: mechanical ventilation

INTERVENTIONS:
Device: mechanical ventilation — Connection to mechanical ventilator

SUMMARY:
Hospital-acquired pneumonia (HAP) in patients in intensive care often requires the mechanical ventilation (MV). Management and weaning from MV are given by specificity of this type of pulmonary inflammation. Enrolled in the retrospective, observational study were all patients older than 18 years staying at the ICU of University Hospital in Olomouc, between 1 January 2011 and 31 December 2016. The determination of the parameters of the MV, ICU length of stay, hospital length of stay and mortality in HAP group were compared with the control group of patients without HAP.

DETAILED DESCRIPTION:
Hospital-acquired pneumonia (HAP) development influences the parameters of mechanical ventilation, intensive care unit (ICU) length of stay, hospital length of stay, need of tracheostomy, bronchoscopy, reconnection to MV and mortality. We respect HAP definition: acute inflammation of the respiratory bronchioles, alveolar structures and pulmonary interstitium. Clinically it is defined as the presence of newly developed or progressive infiltrates on chest radiographs plus at least two other signs of respiratory tract infection: temperature >38 °C, chest pain, purulent sputum, leukocytosis or leukopenia, signs of inflammation on auscultation, cough and/or respiratory insufficiency. HAP is defined as pneumonia that occurs 48 hours or more after admission, which was not incubating at the time of admission. A retrospective, observational study processing data on all consecutive intensive care patients older than 18 years of age between 1 January 2011 and 31 December 2015. The aim was to determine the incidence of potential risk factors and their impact on the development of HAP. The primary outcome was investigation of the relationship between mechanical ventilation parameters and the presence of early- and late-onset HAP. Enrolled in the study were patients staying at the ICU of the Department of Anesthesiology and Intensive Care Medicine, Faculty of Medicine and Dentistry, Palacky University Olomouc and University Hospital Olomouc, between 1 January 2011 and 31 December 2016. The participants were all patients older than 18 years of age consecutively admitted to the ICU.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+
* Need of Mechanical ventilation (Pressure controlled mechanical ventilation or Pressure support ventilation)

Exclusion Criteria:

* Organ donor
* Need Volume controlled mechanical ventilation
* no mechanical ventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Enrolled in the study were patients staying at the ICU of the Department of Anesthesiology and Intensive Care Medicine, Faculty of Medicine and Dentistry, Palacky University Olomouc and University Hospital Olomouc, between 1 January 2011 and 31 December 2015. The participants were all patients older than 18 years of age consecutively admitted to the ICU, who met HAP criteria.
Sampling Method: Probability Sample
Enrollment: 2654 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-04-06 (Actual)

PRIMARY OUTCOMES:
length of mechanical ventilation | during MV
  days of MV

SECONDARY OUTCOMES:
ICU length of stay | 1 month
  length of stay in ICU
Hospital length of stay (LOS) | 1 month
  length of hospital stay
Mortality | 1 month
  mortality during Hospital LOS

OTHER OUTCOMES:
Inspiratory pressure | during MV
  most high inspiratory pressure during MV
Positive end expiratory pressure (PEEP) | during MV
  most high PEEP during MV

CONTACTS AND LOCATIONS:
Overall Officials: Radovan Uvizl, Principal Investigator — UH Olomouc

IPD SHARING:
Plan to Share IPD: No